CLINICAL TRIAL: NCT01350479
Title: Gown and Glove Use to Prevent the Spread of Infection in VA Community Living Centers
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 10-154
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: Cross infection; Long term care
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Swabs of the gowns and gloves of health care workers that interact with the participants will be tested for MRSA and other types of bacteria. Swabs from body sites (e.g. nose) of participants will be tested for MRSA and other types of bacteria.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MRSA colonized: Residents with history of MRSA in the past year
- Not MRSA colonized: Residents without history of MRSA in the past year

SUMMARY:
Methicillin-resistant S. aureus (MRSA) infections are a common cause of morbidity and mortality in nursing home residents. MRSA is predominantly spread from patient-to-patient by health care workers. The use of gowns, gloves and hand washing prevents this spread; however, their use detracts from a patient-centered, home-like environment which is an important priority for nursing homes. The goal of this project is to determine when it is most important for health care workers to wear gowns and to wash their hands when caring for MRSA colonized Veterans in community living centers.

DETAILED DESCRIPTION:
Methicillin-resistant S. aureus (MRSA) infections are a common cause of morbidity and mortality in nursing home residents. MRSA is predominantly spread from patient-to-patient by health care workers. The use of gowns, gloves and hand washing prevents this spread; however, their use detracts from a patient-centered, home-like environment which is an important priority for nursing homes. The goal of this project is to determine when it is most important for health care workers to wear gowns and to wash their hands when caring for MRSA colonized Veterans in community living centers. To meet this goal, the investigators will enroll ~400 MRSA-colonized residents and health care workers from VA community living centers in four states and the District of Columbia. Additionally, the investigators will enroll some non-MRSA colonized residents as control subjects. Each enrolled resident will be followed for 6-25 episodes of care observations over 30 days. During each observation, the investigators will have health care workers wear disposable gowns and gloves during each care activity (e.g. wound dressing) that occurs during the study visit. At the end of each care activity, the investigators will swab the gown and gloves prior to disposing of them. Each swab will be tested for MRSA to determine if MRSA from the resident was transferred to the healthcare worker's gown or gloves during that episode of care. The results of the investigators' analysis will be used to develop new infection control guidelines which balance patient safety and a home-like, patient-centered environment.

ELIGIBILITY:
Inclusion Criteria:

Resident:

* Age 18 years
* Reside in a participating LTCF for rehabilitation, skilled nursing or maintenance care
* Expected length of stay of >4 weeks from enrollment
* Written informed consent from participant, or written informed consent from legally authorized representative (LAR) with assent from participant

Health Care Worker:

* Has direct interaction with participating residents at participating VA Long Term Care Facility (LTCF)
* Verbal informed consent

Exclusion Criteria:

Residents:

* None

Health Care Worker:

* Unable or unwilling to wear protective gown or gloves during healthcare workers (HCW)-resident interaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans residing in a participating VA Long Term Care Facility
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Claire Roghmann, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (7):
- United States (7):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Rehabilitation R&D Service, Baltimore, MD, Baltimore, Maryland
  - Perry Point VA Medical Center VA Maryland Health Care System, Perry Point, MD, Perry Point, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pineles L, Morgan DJ, Lydecker A, Johnson JK, Sorkin JD, Langenberg P, Blanco N, Lesse A, Sellick J, Gupta K, Leykum L, Cadena J, Lepcha N, Roghmann MC. Transmission of methicillin-resistant Staphylococcus aureus to health care worker gowns and gloves during care of residents in Veterans Affairs nursing homes. Am J Infect Control. 2017 Sep 1;45(9):947-953. doi: 10.1016/j.ajic.2017.03.004. Epub 2017 Apr 18. PMID 28431853
- [Derived] Jackson SS, Lydecker AD, Magder LS, Roghmann MC. Development and Validation of a Clinical Prediction Rule to Predict Transmission of Methicillin-Resistant Staphylococcus aureus in Nursing Homes. Am J Epidemiol. 2019 Jan 1;188(1):214-221. doi: 10.1093/aje/kwy220. PMID 30351349
- [Derived] Roghmann MC, Andronescu LR, Stucke EM, Johnson JK. Clostridium difficile Colonization of Nursing Home Residents. Infect Control Hosp Epidemiol. 2017 Oct;38(10):1267-1268. doi: 10.1017/ice.2017.172. Epub 2017 Aug 22. No abstract available. PMID 28826425
- [Derived] Blanco N, Pineles L, Lydecker AD, Johnson JK, Sorkin JD, Morgan DJ; VA Gown and Glove Investigators; Roghmann MC. Transmission of Resistant Gram-Negative Bacteria to Health Care Worker Gowns and Gloves during Care of Nursing Home Residents in Veterans Affairs Community Living Centers. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00790-17. doi: 10.1128/AAC.00790-17. Print 2017 Oct. PMID 28717036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants withdrew from the study prior to cultures being obtained and were not assigned to a study group.
Groups:
- MRSA Colonized: Residents colonized with MRSA by culture at study admission
- Not MRSA Colonized: Residents not colonized with MRSA by culture at study admission
Period: Overall Study
Arm/Group | MRSA Colonized | Not MRSA Colonized
Started | 94 | 106
Completed | 94 | 106
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRSA Colonized | Not MRSA Colonized | Total
Number analyzed (Participants) | 94 | 106 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (13) | 70 (13) | 71 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 92 | 100 | 192
Region of Enrollment [Number; unit: participants]
  United States | 94 | 106 | 200

OUTCOME MEASURES:

1. Primary Outcome: MRSA Transmission
Description: Presence of MRSA on gown or gloves worn by enrolled health care worker for research purposes while providing a specific type of care for enrolled resident
Time Frame: Will be measured during 6-25 episodes of care interactions scheduled over the 30 days following resident enrollment
Population: We analyzed the number of gown and glove swabs from HCW interacting with MRSA and non-MRSA colonized residents.
Measure: Number; unit: Proportion of swabs positive for MRSA
Units Other Than Participants: swabs
Groups:
- Swabs From Interactions With MRSA Colonized Residents: Swabs collected from healthcare workers interacting with residents colonized with MRSA by culture on enrollment
- Swabs From Interactions With Not MRSA Colonized Residents: Swabs collected from healthcare workers interacting with residents not colonized with MRSA by culture on enrollment
Arm/Group | Swabs From Interactions With MRSA Colonized Residents | Swabs From Interactions With Not MRSA Colonized Residents
Number analyzed (Participants) | 94 | 106
Number analyzed (swabs) | 1543 | 1462
Proportion of swabs positive for MRSA
  Proportion of glove swabs with MRSA | 0.20 | 0.02
  Proportion of gown swabs with MRSA | 0.11 | 0.01

ADVERSE EVENTS:
Description: Only serious adverse events were collected.
Arm/Group | MRSA Colonized | Not MRSA Colonized
Serious Adverse Events (participants affected / at risk) | 9/94 | 8/106
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRSA Colonized (N=94) | Not MRSA Colonized (N=106)
Hospitalization (General disorders) | 9 | 6 — Residents transferred from nursing home to acute care hospital, unrelated to study
Death (General disorders) | 0 | 2 — Death of resident unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes